CLINICAL TRIAL: NCT03367585
Title: Effects of Vitamin D Supplementation in Muscle Strength and Postural Balance Training in Vulnerable Elderly Women
Brief Title: Effects of Vitamin D Supplementation in Muscle Strength and Balance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 306/15
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2019-10

CONDITIONS: Osteoporosis, Osteopenia; Osteoporosis, Postmenopausal
Keywords: Supplementary Feeding; vitamin D; Muscle Strength; postural balance; exercise; aged
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Osteoporosis, Postmenopausal; Motor Activity | interventions — Exercise; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Randomized prospective clinical trial, double-blind, placebo-controlled intervention
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group, which will supplement vitamin D3 50,000 IU / week, being in two capsules (25,000 IU / week each),
  Interventions: Dietary Supplement: Physical exercise + Vitamin D3
- Placebo (Placebo Comparator): The placebo group will inject two capsules of equal size, volume and coloration, composed of lactose, without the vitamin D3 supplement.
  Interventions: Other: Physical exercise

INTERVENTIONS:
Dietary Supplement: Physical exercise + Vitamin D3 — Strength exercise + Supplementation of vitamin D3 50,000 IU / week
  Arms: Experimental
Other: Physical exercise — Strength exercise
  Arms: Placebo

SUMMARY:
Introduction: In Brazil, a person who is sixty years old or more is considered elderly. The incidence of osteoporosis and osteopenia has been increasing, as have fractures resulting from falls. Vitamin D deficiency can cause muscular atrophy in type II fibers (fast contraction and strength), which can increase the risk of falls. The aging process produces reduction in the ability of postural control system to maintain postural balance, which may increase postural instability and consequently increase the elderly risk to falls. Objective: To evaluate if vitamin D supplementation associated with regular exercise in vulnerable older women improves muscle strength and postural balance in 12 weeks. Methods: This will be a randomized prospective clinical trial, double blind, placebo-controlled intervention. Will be part of the study 40 elderly women vulnerable, who meet the inclusion criteria and that will be coming from the community through calls made by radio and social network. The volunteer will undergoing to blood test, body composition and bone mineral density, Mini Mental State Examination, Geriatric Depressive Scale, Falls Efficacy Scale, WHOQOL-OLD and WHOQOL-BREF instruments, functional capacity tests (MiniBEST, Time up and Go, Chair Rising Test, Six-minute walk test), muscular strength assessment (isokinetic dynamometry, handgrip and 1RM test) and postural balance (AccSway force platform for static postural balance and NeuroCom's Balance Master for dynamic postural balance) before and after 12 weeks of intervention with vitamin D supplementation and resistance and postural balance exercise. The intervention that will be perform during the 12 weeks with a progressive resistance training program.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 60 years;
2. Osteoporosis or osteopenia (bone mineral density lower than -1.5 standard deviations of the T-score);
3. Present hypovitaminosis D (<30 nmol / L);
4. Do not practice regular resistance exercise;
5. Can not have an injury in lower limbs at least on the last three months,;
6. Be able to perform independent gait without climbing for at least 100 meters;
7. Be independent in your daily life activities;
8. Do not present restrictions for the practice of resistance exercises, including having performed a recent exercise test (maximum 6 months);
9. Do not use medications such as estrogen's, diuretics, to improve bone mass;
10. Do not use dietary supplements with vitamin D;
11. Do not present hyperparathyroidism, diabetes, uncontrolled hypertension, hyperprolactinemia, hypercalciuria, renal lithiasis or elevated serum calcium.

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Postural balance - semi static - change | This measure will be performing before; after the innervation (12 weeks strength and postural balance exercise) and six months after the intervention (six months follow up).
  Evaluation of postural balance - AccSway force platform for semi static postural. The arithmetic mean of the results was calculated from the three tests conducted under each condition, and was processed using the Balance Clinic software. The following parameters were used to measure the stability of the participants: medial-lateral and anteroposterior amplitude (cm), the mean velocity calculated from the total displacement of the center of pressure (COP) in all directions (cm/s), and the elliptical area encompassing 95% of the displacement from the COP (cm2). The following parameters were used to measure the stability of the participants: medial-lateral and anteroposterior amplitude (cm), the mean velocity calculated from the total displacement of the center of pressure (COP) in all directions (cm/s).

SECONDARY OUTCOMES:
Postural balance - dynamic - change | This measure will be performing before; after the innervation (12 weeks strength and postural balance exercise) and six months after the intervention (six months follow up).
  Evaluation of dynamic postural balance - The postural balance assessment (posturography) will be perform on the NeuroCom Balance Master® force platform system (NeuroCom International, Inc., Clackamas, OR, USA). The variables will be the mean sway speed (cm/s) on a stable surface and an unstable surface; and the mean sway in the anteropoterior direction and mediolateral (cm) direction at the same conditions. The variables will be the mean weight transfer index (%), mean movement time (s) and mean impact index.
Muscular strength - Hand Grip - change | This measure will be perform before and after the intervation (12 weeks strenght and potural balance exercise).
  Evaluation of muscular strength improvement- hand grip strength (HGS). HGS assessment was performed using a Jamar hand dynamometer, measured in kilograms (kg), which is adopted by the American Society of Hand Therapists (ASHT).
Muscular strength - Isokinetic dynamometry - change | This measure will be performing before; after the innervation (12 weeks strength and postural balance exercise) and six months after the intervention (six months follow up).
  Evaluation of muscular strength improvement - Isokinetic dynamometry will be use to determine knee extension and flexion strength using the Biodex Multi-Joint System 3 (Biodex MedicalTM, Shirley, NY, USA). The isokinetic variables used were maximum peak torque corrected for body weight (%), and total work (J).
Muscular strength - 1 maximal repetition (RM)- change | This measure will be performing before; after the innervation (12 weeks strength and postural balance exercise) and six months after the intervention (six months follow up).
  Evaluation of muscular strength improvement - 1RM test. One-repetition maximum in weight training is the maximum amount of force that can be generated in one maximal contraction (kg).
Body composition and bone mineral density - change | This measure will be performing before; after the innervation (12 weeks strength and postural balance exercise) and six months after the intervention (six months follow up).
  Evaluation of body composition (area=cm2; BMC=g and BMD=g/cm2) and bone mineral density (BMD=g/cm2; T-score)

CONTACTS AND LOCATIONS:
Locations (1):
- Julia Maria DÀndrea Greve, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No